CLINICAL TRIAL: NCT02855268
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, Pharmacodynamics, and Pharmacokinetics of Lademirsen (SAR339375) for Subcutaneous Injection Administered Every Week in Patients With Alport Syndrome
Brief Title: Study of Lademirsen (SAR339375) in Patients With Alport Syndrome
Acronym: HERA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results of the futility analysis led to the study termination. No unexpected safety findings were identified.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT16248; 2019-004394-10 (EudraCT Number)
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Alport Syndrome
Keywords: Kidney disease; Nephritis; Hereditary nephritis; Hereditary kidney disease
MeSH Terms: conditions — Nephritis, Hereditary; Kidney Diseases; Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo/Lademirsen (Experimental): Participants received subcutaneous (SC) doses of placebo (matched to lademirsen) every week (QW) during the 48 weeks of double blind (DB) treatment period. Participants who received placebo and completed DB treatment period entered in open-label extension (OLE) treatment period and received lademirsen at a dose of 110 milligrams (mg) QW for an additional 48 weeks (i.e., up to Week 96).
  Interventions: Drug: lademirsen (SAR339375)
- Lademirsen/Lademirsen (Experimental): Participants received SC doses of lademirsen 110 mg QW during the 48 weeks of DB treatment period. Participants who completed DB treatment period entered in OLE treatment period and continued the same lademirsen treatment in OLE period for an additional 48 weeks (i.e., up to Week 96).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lademirsen (SAR339375) — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous injection
  Arms: Placebo/Lademirsen
Drug: Placebo — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous injection
  Arms: Lademirsen/Lademirsen

SUMMARY:
Primary Objectives:

* To assess the efficacy of lademirsen (SAR339375) in reducing the decline in renal function.
* To assess the safety and tolerability of lademirsen (SAR339375) in participants with Alport syndrome.

Secondary Objectives:

* To assess plasma pharmacokinetic (PK) parameters of the parent compound and its active major metabolite.
* To assess the potential formation of anti-drug antibodies (ADAs) following administration of lademirsen (SAR339375).
* To assess the pharmacodynamic effect of lademirsen (SAR339375) on miR-21 and on changes in renal injury and function biomarkers.

DETAILED DESCRIPTION:
The planned length of participation in the study for each participant was up to approximately 110 weeks (from screening through completion of follow-up). This included:

* Screening/baseline period of up to 4 weeks
* Double-blind, placebo-controlled treatment period of 48 weeks
* Open-label extension treatment period of 48 weeks (all participant to enter a 48-week open label extension period and receive active treatment with lademirsen [SAR339375]).
* Post-treatment follow-up period of 10 weeks.

ELIGIBILITY:
Inclusion criteria:

* Male or female.
* Confirmed diagnosis of Alport syndrome

  1. Clinical diagnosis (hematuria, family history, hearing loss, ocular change), AND
  2. Genetic confirmation of Alport Syndrome in the participant or the family member, OR
  3. Kidney biopsy showing glomerular basement membrane abnormalities (e.g., significant thinning, thickening, irregularity or lucencies) consistent with Alport Syndrome.
* Age 18-55 years old.
* eGFR > 35 ml/min/1.73m^2 and <90 mL/min/1.73m^2 (based on CKD-EPI) at screening.
* Renal Function Criteria (participants must have met at least one of the following CRITERIA A, B or C):

  * A) Decline in eGFR of >=4 mL/min/1.73 m^2/year (eGFR slope <= -4) based on a linear regression slope analysis of >=4 eGFR measurements within 3 years prior to the study and with a minimum of 2-year time span (the last, of the screening measurement, and first eGFR measurements should be separated by at least 2 years). eGFR was calculated by using either the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation.
  * B) proteinuria (UPCR) >2000 mg/g (UACR>1000 mg/g).
  * C) Age and sex adjusted eGFR (based on CKD-Epi; male 18-23 eGFR<90 mL/min/1.73m^2
* ACE inhibitor and/or ARB, the dosing regimen should be stable for at least 30 days prior to screening.
* Sexually active female participants of childbearing potential and sexually mature male participants must have agreed to practice true abstinence in line with their preferred and usual lifestyle or to use two acceptable effective methods of contraception for the entire duration of the study and for at least 6 weeks after last dose.
* Negative drug screen for opiates, cocaine, heroin, phencyclidine, amphetamines (including ecstasy), barbiturates, benzodiazepines, and cannabinoids. At the Investigator's discretion, participants prescribed benzodiazepines, cannabinoids, or opiates with positive results on a drug screen were allowed.
* Negative screening results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
* Normal biological tests.
* Able to understand all study procedures in the informed consent form (ICF) and to comply with all aspects of the protocol.

Exclusion criteria:

* Causes of chronic kidney disease aside from Alport syndrome (including but not limited to other heritable disorders leading to chronic kidney disease, diabetic nephropathy, hypertensive nephropathy, lupus nephritis, IgA nephropathy).
* End stage renal disease (ESRD) as evidenced by ongoing dialysis therapy or history of renal transplantation.
* Any clinically significant illness within 30 days before screening or surgical or medical condition (other than Alport syndrome) that could interfere with the participant's study compliance; confound the study results; impact participant safety; or significantly alter the absorption, distribution, metabolism, or excretion of drugs.
* Weight > 110 kg.
* Any history of active malignancy within the last 1 year (history of localized basal cell or squamous cell carcinoma and cervical carcinoma in situ that has been excised/appropriately treated or a fully excised malignant lesion with a low probability of recurrence will not be considered exclusionary).
* Prior treatment with Bardoxolone within 90 days prior to screening.
* History or presence of alcoholism or drug abuse within 2 years before screening or other concurrent social conditions that would potentially interfere with the participant's study compliance, at the discretion of the Investigator.
* Participation in a recent investigational study and receipt of an investigational drug or investigational use of a licensed drug within 30 days or 5 half-lives, whichever was longer, prior to screening.
* History or presence of hypersensitivity or idiosyncratic, allergic, or other clinically significant reaction to the study drug (including placebo), inactive ingredients, or related compounds (e.g., other oligonucleotide products).
* Any other condition or circumstance that, in the opinion of the Investigator, may make the participant unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the participant's safety and well-being.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- United States (5):
  - Investigational Site Number :8400002, Los Angeles, California
  - University of Minnesota Childrens' Hospital_Investigational Site Number :8400003, Minneapolis, Minnesota
  - Columbia University Medical Center_Investigational Site Number :8400004, New York, New York
  - The Cleveland Clinic Foundation_Investigational Site Number :8400001, Cleveland, Ohio
  - University of Utah_Investigational Site Number :8400005, Salt Lake City, Utah
- Australia (3):
  - Investigational Site Number :0360003, Herston, Queensland
  - Investigational Site Number :0360001, Parkville, Victoria
  - Investigational Site Number :0360002, Nedlands, Western Australia
- China (3):
  - Investigational Site Number :1560001, Beijing
  - Investigational Site Number :1560002, Beijing
  - Investigational Site Number :1560004, Guangzhou
- France (2):
  - Investigational Site Number :2500001, Paris
  - Investigational Site Number :2500002, Toulouse
- Germany (2):
  - Uniklinik Köln, Innere Medizin II - Nephrologie, Rheumatologie, Diabetologie und Allgemeine Innere Medizin_Investigational Site Number :2760001, Cologne
  - Universitätsmedizin Göttingen, Klinik für Nephrologie und Rheumatologie_Investigational Site Number :2760002, Göttingen
- Spain (5):
  - Investigational Site Number :7240005, Córdoba, Andalusia
  - Investigational Site Number :7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240002, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240003, Granada
- United Kingdom (3):
  - Investigational Site Number :8260001, London, London, City of
  - Investigational Site Number :8260002, Nottingham, Nottinghamshire
  - Investigational Site Number :8260003, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gale DP, Gross O, Wang F, Esteban de la Rosa RJ, Hall M, Sayer JA, Appel G, Hariri A, Liu S, Maski M, Shen Y, Zhang Q, Iqbal S, Kowthalam MU, Lin J, Ding J; HERA Clinical Trial Group. A Randomized Controlled Clinical Trial Testing Effects of Lademirsen on Kidney Function Decline in Adults with Alport Syndrome. Clin J Am Soc Nephrol. 2024 Aug 1;19(8):995-1004. doi: 10.2215/CJN.0000000000000458. Epub 2024 Jun 3. PMID 38829703
- [Derived] Kashtan CE, Gross O. Clinical practice recommendations for the diagnosis and management of Alport syndrome in children, adolescents, and young adults-an update for 2020. Pediatr Nephrol. 2021 Mar;36(3):711-719. doi: 10.1007/s00467-020-04819-6. Epub 2020 Nov 6. PMID 33159213
- See also: ACT16248 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25190&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 active centers in 7 countries. A total of 67 participants were screened between 02 November 2019 and 30 December 2021, out of which 43 participants were randomized.
Pre-assignment Details: The study was planned with 2 Stages/Cohorts. Since the study was terminated early, Stage 2/Cohort 2 was not conducted. In Stage 1 analysis of double blind (DB) period performed until 48 weeks. In Stage 1 open label extension (OLE) period, only safety data was collected and assessed due to early study termination.
Groups:
- Placebo/Lademirsen: Participants received subcutaneous (SC) doses of placebo (matched to lademirsen) every week (QW) during the 48 weeks of DB treatment period. Participants who received placebo and completed DB treatment period entered in OLE treatment period and received lademirsen at a dose of 110 milligrams (mg) QW for an additional 48 weeks (i.e., up to Week 96).
Period: DB Period (up to 48 Weeks)
Arm/Group | Placebo/Lademirsen | Lademirsen/Lademirsen
Started | 14 | 29
Completed | 9 | 19
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Sponsor Decision | 4 | 7
Period: OLE Period (up to 96 Weeks)
Arm/Group | Placebo/Lademirsen | Lademirsen/Lademirsen
Started | 9 | 19
Completed | 1 | 0
Not Completed | 8 | 19
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Early study termination by sponsor | 7 | 16

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized population.
Groups:
- Placebo/Lademirsen: Participants received SC doses of placebo (matched to lademirsen) QW during the 48 weeks of DB treatment period. Participants who received placebo and completed DB treatment period entered in OLE treatment period and received lademirsen at a dose of 110 mg QW for an additional 48 weeks (i.e., up to Week 96).
- Total: Total of all reporting groups
Arm/Group | Placebo/Lademirsen | Lademirsen/Lademirsen | Total
Number analyzed (Participants) | 14 | 29 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (12.0) | 34.5 (11.5) | 33.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 7 | 19 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 19 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
eGFR value [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR was used to measure level of kidney function and determine the stage of kidney disease. eGFR was calculated using CKD-EPI Creatinine Equation as: eGFR =142*min (Scr/K, 1) α*max (Scr/K, 1)^-1.200*0.9938^Age*1.012 [if female], where Scr was serum creatinine in mg/dL, K is 0.7 for females and 0.9 for males, α was -0.241 for females and -0.302 for males. age=years, calculated at time of creatinine measurement.
  mL/min/1.73m^2 | 57.397 (16.514) | 54.801 (15.726) | 55.646 (15.837)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE): any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs: AEs with onset after the first dose of investigational medicinal product (IMP) or existing AEs that worsened during TEAE Period (for DB Period: from first IMP administration up to first administration in OLE period for participant who entered OLE period; and up to 7 days post last IMP administration for participant not continuing OLE period; for open-label: time from 1st IMP administration in open-label to last IMP administration+ 10 weeks).
Time Frame: DB: from 1st dose of IMP upto 1st dose of IMP in OLE for participant who entered OLE (Week 48); up to 7 days post last dose for participant not continuing to OLE (Week 49); OLE:1st dose of IMP (at Week 48) in OLE upto 10 weeks post last dose (Week 106)
Population: Analysis was performed on safety population that included all participants who received at least one dose or partial of a dose of the IMP, analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Groups:
- DB Period: Placebo: Participants received SC doses of placebo (matched to lademirsen) QW during the 48 weeks of DB treatment period.
- DB Period: Lademirsen: Participants received SC doses of lademirsen 110 mg QW during the 48 weeks of DB treatment period.
- OLE Period: Placebo/Lademirsen: Participants who completed DB treatment period with placebo (matched to lademirsen) QW, entered in OLE treatment period and received lademirsen at a dose of 110 mg QW for an additional 48 weeks (i.e., up to Week 96).
- OLE Period: Lademirsen/Lademirsen: Participants who completed DB treatment period with lademirsen 110 mg QW, entered in OLE treatment period and continued the same lademirsen treatment in OLE period for an additional 48 weeks (i.e., up to Week 96).
Arm/Group | DB Period: Placebo | DB Period: Lademirsen | OLE Period: Placebo/Lademirsen | OLE Period: Lademirsen/Lademirsen
Number analyzed (Participants) | 14 | 29 | 9 | 19
Participants
  TEAE | 14 | 29 | 8 | 19
  TESAE | 0 | 2 | 2 | 1

2. Primary Outcome: DB Period: Annualized Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 48
Description: Annualized change in eGFR was calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation (for participants with age greater than 16 years) as: eGFR=142*min(Scr/K, 1)α*max(Scr/K, 1)^-1.200*0.9938^Age*1.012 [if female], where Scr = serum creatinine in milligrams per deciliter (mg/dL), K = 0.7 for females (F) and 0.9 for males (M), α = -0.241(F) and -0.302(M); age=years, calculated at time of creatinine measurement. eGFR measurements collected from baseline to Week 48 were the response variable and included fixed effects of treatment (lademirsen or placebo), screening eGFR stratification factor (less than [<]60 versus greater than or equal to [>=]60 milliliters per minute per 1.73 meters squared [mL/min/1.73 m^2]), time, and treatment-by-time interaction. Least square (LS) mean and standard error (SE) estimated by linear mixed effect model.
Time Frame: Baseline, Week 48
Population: Analysis was performed on primary population that included all randomized participants who completed the double-blinded period (the first 48 weeks) or discontinued double-blinded period early.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2/year
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 10 | 20
mL/min/1.73 m^2/year | -4.70 (2.69) | -4.91 (1.86)
Statistical Analysis 1: Comparison: DB Period: Placebo vs DB Period: Lademirsen; Annualized rate of change in eGFR during the placebo-controlled treatment period was compared between lademirsen and placebo using a random coefficient linear mixed effect model which included time as a continuous variable; Test type: Superiority; p = 0.9472, Linear mixed effect model — Threshold of significance was 1-sided <0.025; Least square mean difference = -0.22, 95% CI 2-sided [-6.92 to 6.48], Standard Error of Mean 3.27

3. Secondary Outcome: DB Period: Absolute Change From Baseline in eGFR Values at Week 24 and 48
Description: eGFR was used to measure level of kidney function and determine the stage of kidney disease. eGFR was calculated using CKD-EPI Creatinine Equation as: eGFR =142*min (Scr/K, 1) α*max (Scr/K, 1)^-1.200*0.9938^Age*1.012 [if female], where Scr was serum creatinine in mg/dL, K is 0.7 for females and 0.9 for males, α was -0.241 for females and -0.302 for males. Unit of age was years, calculated to reflect the age at the time when creatinine was measured.
Time Frame: Baseline, Weeks 24 and 48
Population: Analysis was performed on Intent-to-Treat (ITT) population that included all randomized participants analyzed according to the treatment group allocated by randomization. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
mL/min/1.73 m^2
  Week 24 | -3.43 (2.74) | -5.15 (1.84)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | -7.08 (3.00) | -6.89 (2.02)

4. Secondary Outcome: DB Period: Percent Change From Baseline in eGFR Values at Week 24 and 48
Description: as for outcome 3
Time Frame: Baseline, Weeks 24 and 48
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
percent change
  Week 24 | -4.78 (4.51) | -8.44 (3.03)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | -10.05 (5.64) | -12.77 (3.79)

5. Secondary Outcome: DB Period: Number of Participants With a Reduction From Baseline in eGFR of <10%, <20%, <30%, or <40% at Weeks 24 and 48
Description: Estimated glomerular filtration rate was used to measure level of kidney function and determine the stage of kidney disease. eGFR was calculated using CKD-EPI Creatinine Equation as: eGFR = 142*min(Scr/K,1)α*max(Scr/K,1)^-1.200*0.9938^Age*1.012 [if female], where Scr was serum creatinine in mg/dL, K is 0.7 for females and 0.9 for males, α was -0.241 for females and -0.302 for males. Number of participants with a reduction from baseline in eGFR value of <10%, <20%, <30%, or <40% at Weeks 24 and 48 were reported in this outcome measure.
Time Frame: At Weeks 24 and 48
Population: Analysis was performed on ITT population. Here, 'number analyzed' = participants considered for the analysis for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  <10% reduction: Week 24 | 7 | 16
  <20% reduction: Week 24 | 11 | 23
  <30% reduction: Week 24 | 12 | 26
  <40% reduction: Week 24 | 12 | 26
  <10% reduction: Week 48: number analyzed (Participants) | 10 | 20
  <10% reduction: Week 48 | 5 | 8
  <20% reduction: Week 48: number analyzed (Participants) | 10 | 20
  <20% reduction: Week 48 | 7 | 13
  <30% reduction: Week 48: number analyzed (Participants) | 10 | 20
  <30% reduction: Week 48 | 9 | 14
  <40% reduction: Week 48: number analyzed (Participants) | 10 | 20
  <40% reduction: Week 48 | 9 | 16

6. Secondary Outcome: DB Period: Number of Participants Who Developed End Stage Renal Disease (ESRD)
Description: ESRD was defined as: eGFR <=15 mL/min/1.73 m^2; or initiation of hemodialysis; or receiving a renal transplantation during the double-blind treatment period.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants | 0 | 1

7. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities (PCSA): Hematological Parameters
Description: Criteria for PCSA included: Hemoglobin (Hb): <= 115 grams per liter (g/L) (Male), <= 95 g/L (Female); greater than or equal to (>=) 185 g/L (18.5 g/dL) (Male), >= 165 g/L (16.5g/dL) (Female); decrease from Baseline (DFB) = 20 g/L (2g/dL); Hematocrit: <= 0.37 volume/volume (v/v) (Male); <= 0.32 v/v (Female); >= 0.55 v/v (Male); >= 0.5 v/v (Female); Red Blood Cells (RBCs):>=6 Tera/ liter (L) and Platelets: <100 Giga/L; >= 700 Giga/L.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  Hb:<=115 g/L, <=95 g/L | 4 | 5
  Hb: >=185 g/L, >=165 g/L | 0 | 0
  Hb: DFB >=20 g/L | 1 | 2
  Hematocrit: <= 0.37 v/v; <=0.32 v/v | 9 | 18
  Hematocrit: >=0.55 v/v; >=0.5 v/v | 0 | 0
  RBCs: >=6 Tera/L | 0 | 0
  Platelets: <100 Giga/L | 0 | 0
  Platelets: >= 700 Giga/L | 0 | 0

8. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for potentially clinically significant abnormalities: Creatinine: >=150 micromol/L (adults); >=30% change from baseline, >=100% change from baseline; Blood urea nitrogen: >=17 millimoles per liter (mmol/L); Uric acid: <120 micromol/L; >408 micromol/L; Creatinine clearance: <15 mL/min; >=15 to <30 mL/min; >=30 to <60 mL/min; >=60 to <90 mL/min; >=90 mL/min; eGFR: < 15 mL/min/1.73m^2; >=15 to <30 mL/min/1.73m^2; >=30 to <60 mL/min/1.73m^2; >=60 to <90 mL/min/1.73m^2; >=90 mL/min. Participants might be counted more than once for specified categories.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  Creatinine >=150 micromol/L | 9 | 21
  Creatinine >=30%change from baseline | 3 | 13
  Creatinine >=100% change from baseline | 0 | 2
  Blood urea nitrogen: >=17 mmol/L | 2 | 9
  Uric acid <120 micromol/L | 0 | 0
  Uric acid >408 micromol/L | 13 | 22
  Creatinine clearance <15 mL/min | 0 | 1
  Creatinine clearance >=15 to <30mL/min | 2 | 4
  Creatinine clearance >=30 to <60 mL/min | 8 | 21
  Creatinine clearance >=60 to <90 mL/min | 7 | 17
  Creatinine clearance >=90 mL/min | 2 | 5
  eGFR <15 mL/min/1.73m^2 | 0 | 1
  eGFR >=15 to <30 mL/min/1.73m^2 | 0 | 5
  eGFR >=30 to <60 mL/min/1.73m^2 | 12 | 26
  eGFR >=60 to <90 mL/min/1.73m^2 | 6 | 11
  eGFR >=90 mL/min | 1 | 3

9. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for PCSA: Total bilirubin (TBILI): >1.5 upper limit of normal (ULN); >2 ULN; Alanine Aminotransferase (ALT): >3 ULN; >5 ULN; >10 ULN; >20 ULN; Aspartate aminotransferase (AST): >3ULN; >5 ULN; >10 ULN; >20 ULN; Alkaline phosphatase: >1.5 ULN; ALT>3 ULN and TBILI>2 ULN and Direct Bilirubin> 35% TBILI and TBILI> 1.5 ULN.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  TBILI >1.5 ULN | 0 | 0
  TBILI >2 ULN | 0 | 0
  ALT >3 ULN | 0 | 0
  ALT >5 ULN | 0 | 0
  ALT >10 ULN | 0 | 0
  ALT >20 ULN | 0 | 0
  AST >3 ULN | 0 | 0
  AST >5 ULN | 0 | 0
  AST >10 ULN | 0 | 0
  AST >20 ULN | 0 | 0
  ALP >1.5 ULN | 0 | 0
  ALT >3 ULN and TBILI >2 ULN | 0 | 0
  Direct Bilirubin >35% TBILI and TBILI >1.5 ULN | 0 | 0

10. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Criteria for potentially clinically significant vital sign abnormalities: Systolic blood pressure (SBP):<=95 mmHg and DFB >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg; SBP (Orthostatic): <=-20mmHg; Diastolic blood pressure (DBP): <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg; DBP (Orthostatic): <=10 mmHg; heart rate (HR): <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB>=20 bpm and Weight: >=5% DFB; >=5% IFB.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  SBP <=95 mmHg and DFB >=20 mmHg | 0 | 1
  SBP >=160 mmHg and IFB >=20 mmHg | 0 | 2
  SBP (Orthostatic) <=-20mmHg | 0 | 0
  DBP <=45 mmHg and DFB >=10 mmHg | 0 | 0
  DBP >=110 mmHg and IFB >=10 mmHg | 0 | 0
  DBP (Orthostatic) <=-10 mmHg | 0 | 0
  HR <=50 bpm and DFB >=20 bpm | 0 | 0
  HR >=120 bpm and IFB>=20 bpm | 0 | 0
  Weight >=5% DFB | 1 | 3
  Weight >=5% IFB | 4 | 4

11. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) Findings
Description: Criteria for potentially clinically significant ECG abnormalities: HR: <50 bpm; <50 bpm and DFB >=20 bpm; <40 bpm; <40 bpm and DFB >=20 bpm; <30 bpm; <30 bpm and DFB >=20 bpm; >90 bpm; >=90 bpm and IFB >=20 bpm; >100 bpm; >=100bpm and IFB >=20 bpm; >120 bpm; >=120 bpm and IFB >=20 bpm; PR Interval: >200 millisecond(ms); >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB>=25%; QRS Interval: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%; QT Interval: >500 ms and QTc Fridericia (QTc F): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms.
Time Frame: From Baseline up to Week 48
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 14 | 29
Participants
  HR <50 bpm | 2 | 3
  HR <50 bpm and DFB >=20 bpm | 0 | 0
  HR <40 bpm | 0 | 0
  HR <40 bpm and DFB >=20 bpm | 0 | 0
  HR <30 bpm | 0 | 0
  HR <30 bpm and DFB >=20 bpm | 0 | 0
  HR >90 bpm | 1 | 1
  HR >=90 bpm and IFB >=20 bpm | 0 | 0
  HR >100 bpm | 1 | 1
  HR >=100 bpm and IFB >=20 bpm | 0 | 0
  HR >120 bpm | 0 | 0
  HR >=120 bpm and IFB >=20 bpm | 0 | 0
  PR >200 ms | 0 | 1
  PR >200 ms and IFB >=25% | 0 | 0
  PR >220 ms | 0 | 0
  PR >220 ms and IFB >=25% | 0 | 0
  PR >240 ms | 0 | 0
  PR >240 ms and IFB>=25% | 0 | 0
  QRS Interval >110 ms | 0 | 0
  QRS Interval >110 ms and IFB >=25% | 0 | 0
  QRS Interval >120 ms | 0 | 0
  QRS Interval >120 ms and IFB >=25% | 0 | 0
  QT Interval >500 ms | 0 | 0
  QTcF >450 ms | 0 | 0
  QTcF >480 ms | 0 | 0
  QTcF >500 ms | 0 | 0
  QTcF IFB >30 and <=60 ms | 1 | 4
  QTcF IFB >60 ms | 0 | 0

12. Secondary Outcome: DB Period: Pharmacokinetics (PK): Plasma Concentration of Lademirsen, Its Metabolite (RG0005) and SUM (Lademirsen+RG0005)
Description: Post-dose (4 hours) plasma concentration of lademirsen, its active major metabolite (RG0005), and SUM (lademirsen+RG0005) on Day 1, and at Weeks 24 and 48 are reported in the outcome measure. 4-hour SUM concentrations are calculated values (sum of measured lademirsen+RG0005).
Time Frame: Post-dose (4 hours) on Day 1, Weeks 24 and 48
Population: Analysis was performed on PK population that included all participants who received at least one dose of IMP and had at least one post-dose PK sample. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | DB Period: Lademirsen
Number analyzed (Participants) | 21
nanograms per milliliter
  Lademirsen: Day 1 | 2070 (1150)
  Lademirsen: Week 24: number analyzed (Participants) | 14
  Lademirsen: Week 24 | 2180 (976)
  Lademirsen: Week 48: number analyzed (Participants) | 9
  Lademirsen: Week 48 | 3080 (2170)
  RG0005: Day 1 | 765 (524)
  RG0005: Week 24: number analyzed (Participants) | 14
  RG0005: Week 24 | 835 (441)
  RG0005: Week 48: number analyzed (Participants) | 9
  RG0005: Week 48 | 876 (460)
  Lademirsen + RG0005: Day 1 | 2840 (1660)
  Lademirsen + RG0005: Week 24: number analyzed (Participants) | 14
  Lademirsen + RG0005: Week 24 | 3020 (1410)
  Lademirsen + RG0005: Week 48: number analyzed (Participants) | 9
  Lademirsen + RG0005: Week 48 | 3960 (2350)

13. Secondary Outcome: DB Period: Pharmacokinetics: Trough Plasma Concentrations (Ctrough) of SUM (Lademirsen+RG0005)
Description: Ctrough was measured from the pre-dose (up to 4 hours before study drug administration) plasma samples collected at Weeks 4, 12, 24, 36 and 48. SUM concentrations (lademirsen+RG0005) are measured values (assay measures lademirsen+ RG0005).
Time Frame: Pre-dose (up to 4 hours before study drug administration) on Weeks 4, 12, 24, 36 and 48
Population: Analysis was performed on PK population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | DB Period: Lademirsen
Number analyzed (Participants) | 13
nanograms per milliliter
  Week 4 | 7.65 (3.36)
  Week 12: number analyzed (Participants) | 12
  Week 12 | 12.6 (7.05)
  Week 24: number analyzed (Participants) | 11
  Week 24 | 15.1 (8.65)
  Week 36: number analyzed (Participants) | 7
  Week 36 | 18.6 (8.18)
  Week 48: number analyzed (Participants) | 5
  Week 48 | 19.5 (10.2)

14. Secondary Outcome: DB Period: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADAs) Response
Description: ADA responses were categorized as: treatment-induced, and treatment-boosted response. Participant whose ADA status was negative at baseline but positive (ADA titer value >=50) anytime post-baseline or missing at baseline was considered to have treatment-induced ADA. Participant whose ADA status was positive at baseline (pre-existing ADA) and the ADA titer level anytime post-baseline was significantly higher (>= twice the minimum required dilution) than that at baseline was considered to have treatment-boosted ADA.
Time Frame: From first IMP administration (Day 1) up to first administration in OLE period for participant who entered OLE period (i.e., up to W48) & up to 7 days post last IMP administration for participant not continuing OLE period (i.e., up to W49)
Population: Analysis was performed on ADA population that included all randomized participants who received at least one dose of study drugs and had at least one post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 11 | 22
Participants
  Treatment-induced ADAs | 0 | 6
  Treatment-boosted ADAs | 0 | 0

15. Secondary Outcome: DB Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Associated With Anti-drug Antibody (ADA) Responses
Description: TEAEs: AE developed/worsened/became serious during TEAE period (from first IMP administration in DB period to first administration in OLE period for those who entered OLE (i.e., up to W48), up to 7 days post last dose for those not continuing to OLE period (i.e., up to W49). TESAEs: any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization/prolongation of hospitalization, resulted in persistent/significant disability, was a congenital anomaly/birth defect, or a medically important event. ADA response was categorized as treatment-induced (participant whose ADA status was positive [ADA titer value >=50] anytime post-baseline and was negative/missing at baseline), treatment-boosted (participant whose ADA status was positive at baseline & ADA titer level anytime post-baseline was significantly higher). In this outcome measure, number of participants with TEAEs as per ADA responses (positive or negative) were reported.
Time Frame: as for outcome 14
Population: Analysis was performed on ADA population. For this outcome measure analysis was done separately for TE-ADA positive and negative participants for placebo and lademirsen arms respectively. Here, "0" in the "overall number of participants analyzed" signifies that no participants had ADA positive response in the placebo arm.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: TE-ADA Positive: Participants received SC doses of placebo (matched to lademirsen) QW during the 48 weeks of DB treatment period. ADA positive were participants with treatment induced or treatment boosted ADAs that occurred at any time after the first administration of IMP during the DB treatment period.
- Placebo: TE-ADA Negative: Participants received SC doses of placebo (matched to lademirsen) QW during the 48 weeks of DB treatment period. ADA negative were participants with neither treatment induced nor treatment boosted ADAs at all time after the first administration of IMP during the DB treatment period.
- Lademirsen: TE-ADA Positive: Participants received SC doses of lademirsen 110 mg QW during the 48 weeks of DB treatment period. ADA positive were participants with treatment induced or treatment boosted ADAs that occurred at any time after the first administration of IMP during the DB treatment period.
- Lademirsen: TE-ADA Negative: Participants received SC doses of lademirsen 110 mg QW during the 48 weeks of DB treatment period. ADA negative were participants with neither treatment induced nor treatment boosted ADAs at all time after the first administration of IMP during the DB treatment period.
Arm/Group | Placebo: TE-ADA Positive | Placebo: TE-ADA Negative | Lademirsen: TE-ADA Positive | Lademirsen: TE-ADA Negative
Number analyzed (Participants) | 0 | 11 | 6 | 16
Participants
  TEAEs |  | 11 | 6 | 16
  TESAEs |  | 0 | 0 | 1

16. Secondary Outcome: DB Period: Change From Baseline in Circulating MicroRNA-21 at Weeks 24 and 48
Description: Circulating microRNA-21 were the supportive biomarkers assessed in study.
Time Frame: Baseline, Weeks 24 and 48
Population: Data for this outcome measure could not be analyzed and reported as the samples for circulating microRNA-21 at the predefined timepoints, Weeks 24 and 48 were not collected and analyzed due to early study termination.
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: DB Period: Change From Baseline in Blood Urea Nitrogen (BUN) Values at Weeks 24 and 48
Description: BUN was the supportive biomarker assessed during the study. Change from Baseline in BUN at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
milligrams per deciliter (mg/dL)
  Week 24 | -0.89 (5.96) | 2.54 (8.07)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | -1.54 (7.23) | 5.80 (6.09)

18. Secondary Outcome: DB Period: Change From Baseline in Urine Protein/Creatinine Ratio at Weeks 24 and 48
Description: Urine protein and creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine protein to creatinine ratio at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 11 | 22
ratio
  Week 24 | -0.085 (1.680) | 0.438 (1.451)
  Week 48: number analyzed (Participants) | 7 | 17
  Week 48 | 0.300 (2.308) | 0.745 (1.149)

19. Secondary Outcome: DB Period: Change From Baseline in Urine Albumin/Creatinine Ratio at Weeks 24 and 48
Description: Urine albumin and creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine albumin to creatinine ratio at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 11 | 24
ratio
  Week 24 | 11.65 (1436.63) | 271.28 (1066.40)
  Week 48: number analyzed (Participants) | 8 | 17
  Week 48 | 206.01 (1585.93) | 447.54 (863.94)

20. Secondary Outcome: DB Period: Change From Baseline in Urine Epidermal Growth Factor (EGF)/Creatinine Ratio at Weeks 24 and 48
Description: EGF and creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine EGF to creatinine ratio at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 6 | 19
ratio
  Week 24 | -5.03 (5.42) | 1.84 (7.28)
  Week 48: number analyzed (Participants) | 6 | 13
  Week 48 | -5.48 (7.04) | 0.37 (2.00)

21. Secondary Outcome: DB Period: Change From Baseline in Blood Creatinine Values at Weeks 24 and 48
Description: Creatinine was the supportive biomarker assessed during the study. Change from Baseline in blood creatinine values at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
mg/dL
  Week 24 | 0.082 (0.201) | 0.173 (0.354)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | 0.119 (0.186) | 0.201 (0.403)

22. Secondary Outcome: DB Period: Change From Baseline in Urine Creatinine Values at Weeks 24 and 48
Description: Creatinine was the supportive biomarker assessed during the study. Change from Baseline in urine creatinine values at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 27
mg/dL
  Week 24 | -0.319 (62.960) | -3.595 (38.344)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | -16.461 (55.160) | -24.880 (30.789)

23. Secondary Outcome: DB Period: Change From Baseline in Blood Cystatine C Values at Weeks 24 and 48
Description: Cystatine C was the supportive biomarker assessed during the study. Change from Baseline in blood cystatine C values at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
mg/dL
  Week 24 | 0.061 (0.191) | 0.159 (0.269)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | 0.147 (0.258) | 0.282 (0.387)

24. Secondary Outcome: DB Period: Change From Baseline in Urine Cystatin C/Creatinine Ratio at Weeks 24 and 48
Description: Cystatin C and Creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine cystatin C to creatinine ratio at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 4 | 15
ratio
  Week 24 | 35.203 (146.405) | 201.681 (1030.016)
  Week 48: number analyzed (Participants) | 4 | 9
  Week 48 | 81.309 (106.162) | 41.290 (194.150)

25. Secondary Outcome: DB Period: Change From Baseline in Blood Transforming Growth Factor Beta 1 Values at Week 24 and 48
Description: Transforming growth factor beta 1 was the supportive biomarker assessed during the study. Change from Baseline in blood transforming growth factor beta 1 values at Week 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 5 | 15
nanograms per milliliter (ng/mL)
  Week 24 | 15.66 (19.59) | 0.06 (21.46)
  Week 48: number analyzed (Participants) | 3 | 8
  Week 48 | -5.87 (13.76) | 0.89 (15.08)

26. Secondary Outcome: DB Period: Change From Baseline in Urine Transforming Growth Factor Beta 1/Creatinine Ratio at Week 24 and 48
Description: Transforming growth factor beta 1 and creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine transforming growth factor beta 1 to creatinine ratio at Week 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 6 | 19
ratio
  Week 24 | 6031.03 (13412.10) | 1088.87 (4990.98)
  Week 48: number analyzed (Participants) | 6 | 13
  Week 48 | -636.16 (2864.99) | 1268.16 (6000.78)

27. Secondary Outcome: DB Period: Change From Baseline in Blood Lipocalin-2 Values at Weeks 24 and 48
Description: Blood Lipocalin-2 was the supportive biomarker assessed during the study. Change from Baseline in blood lipocalin-2 at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 12 | 28
micrograms per liter (mcg/L)
  Week 24 | 6.3989 (38.2043) | 14.9748 (62.3959)
  Week 48: number analyzed (Participants) | 9 | 17
  Week 48 | 25.5433 (32.6328) | 31.0391 (41.2171)

28. Secondary Outcome: DB Period: Change From Baseline in Urine Lipocalin-2/Creatinine Ratio at Weeks 24 and 48
Description: Lipocalin-2 and Creatinine were the supportive biomarker assessed during the study. Change from Baseline in urine lipocalin-2 to creatinine ratio at Weeks 24 and 48 was reported in this outcome measure.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DB Period: Placebo | DB Period: Lademirsen
Number analyzed (Participants) | 10 | 26
ratio
  Week 24 | -14.7119 (25.6736) | 16.7727 (173.1358)
  Week 48: number analyzed (Participants) | 8 | 15
  Week 48 | 65.9768 (107.4255) | 47.5224 (101.1673)

ADVERSE EVENTS:
Time Frame: DB period: First IMP administration in DB period up to first IMP administration in OLE period for participant who entered OLE period (i.e., up to Week 48); and up to 7 days post last IMP administration for participant who didn't enter OLE period (i.e., up to Week 49). OLE period: first IMP administration (at Week 48) in OLE period upto 10 weeks post last IMP administration (i.e., up to Week 106)
Description: Analysis was performed on safety population.
Arm/Group | DB Period: Placebo | DB Period: Lademirsen | OLE Period: Placebo/Lademirsen | OLE Period: Lademirsen/Lademirsen
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/29 | 0/9 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/29 | 2/9 | 1/19
Other Adverse Events (participants affected / at risk) | 14/14 | 29/29 | 8/9 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=14) | DB Period: Lademirsen (N=29) | OLE Period: Placebo/Lademirsen (N=9) | OLE Period: Lademirsen/Lademirsen (N=19)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complex Regional Pain Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=14) | DB Period: Lademirsen (N=29) | OLE Period: Placebo/Lademirsen (N=9) | OLE Period: Lademirsen/Lademirsen (N=19)
Covid-19 (Infections and infestations) | 5 (5) | 5 (5) | 1 (1) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis Salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 6 (12) | 1 (3) | 4 (5)
Allergic Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (10) | 3 (10) | 1 (3) | 3 (6)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (12) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 5 (13) | 2 (2) | 3 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 1 (1) | 3 (6)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 4 (5) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (6) | 6 (18) | 0 (0) | 1 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Ophthalmic Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital Swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (6) | 4 (4) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 1 (2) | 0 (0)
Plicated Tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (4) | 3 (3) | 1 (1) | 2 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 2 (2) | 1 (1)
Joint Laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation Delayed (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (7) | 0 (0) | 3 (6)
Fatigue (General disorders) | 2 (3) | 2 (2) | 1 (3) | 1 (1)
Feeling Abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Injection Site Bruising (General disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 1 (1) | 2 (2) | 1 (10) | 1 (1)
Injection Site Haemorrhage (General disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 5 (6) | 2 (2) | 0 (0)
Injection Site Reaction (General disorders) | 6 (14) | 21 (337) | 4 (23) | 9 (88)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Vessel Puncture Site Bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood Bicarbonate Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Parathyroid Hormone Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 10 (18) | 20 (50) | 4 (10) | 8 (11)
Heart Rate Irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sars-Cov-2 Test Positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early study termination, Stage 2/Cohort 2 was not conducted. In Stage 1 analysis of DB period was performed until 48 weeks. In Stage 1 OL period, only safety data was collected and assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02855268/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT02855268/SAP_001.pdf